CLINICAL TRIAL: NCT01959841
Title: Phase III Study of ASP2151 in Herpes Zoster Patients- A Double-blind, Valaciclovir-controlled Study
Brief Title: Phase III Study of ASP2151 in Herpes Zoster Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Maruho Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M522101-J01
Record Dates: First submitted 2013-09-26; First posted 2013-10-10 (Estimated); Results first posted 2018-10-18 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-10

CONDITIONS: Herpes Zoster
MeSH Terms: conditions — Herpes Zoster | interventions — ASP2151; Valacyclovir

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- ASP2151(200 mg) (Experimental): once daily
  Interventions: Drug: ASP2151
- ASP2151(400mg) (Experimental): once daily
  Interventions: Drug: ASP2151
- valaciclovir (Experimental): 1000 mg three times daily
  Interventions: Drug: valaciclovir

INTERVENTIONS:
Drug: ASP2151 — 200 mg once daily or 400 mg once daily
  Arms: ASP2151(200 mg); ASP2151(400mg)
Drug: valaciclovir — 1000 mg three times daily
  Arms: valaciclovir

SUMMARY:
To evaluate the efficacy and safety of ASP2151 (200 mg and 400 mg) in comparison with valaciclovir (VACV) 3000 mg in patients with herpes zoster.

DETAILED DESCRIPTION:
A double-blind, randomized, parallel-group study will be conducted to evaluate the efficacy and safety of ASP2151 (200 mg and 400 mg) in comparison with valaciclovir (VACV) 3000 mg in patients with herpes zoster. The efficacy will be evaluated for the primary endpoint defined as, "the proportion of subjects achieving cessation of new lesion formation by Day 4 of study treatment" to demonstrate the non-inferiority of ASP2151 to VACV. The safety will be evaluated based on adverse events, laboratory tests, vital signs, and ECGs.

ELIGIBILITY:
Inclusion Criteria:

(1) Patients who have a rash associated with herpes zoster, and who can start receiving the study drug within 72 hours after onset of the rash

Exclusion Criteria:

1. Patients who are not expected to have an adequate response to oral antiviral medication
2. An extreme decline in immune function
3. Presence of serious complications
4. Patients found to meet any of the following conditions based on laboratory tests performed within 14 days before informed consent:

   * AST or ALT ≥ 2.5 x upper limit of normal
   * Platelet count < lower limit of normal
   * Serum creatinine ≥ 1.5 mg/dL
   * Creatinine clearance < 50 mL/min
5. Current or previous history of malignant tumor within 5 years before informed consent
6. Diagnosis of autoimmune disease
7. Evidence of bone marrow suppression

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 751 (Actual)
Dates: Start 2013-08; Primary Completion 2015-07 (Actual); Study Completion 2015-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maruho Co.,Ltd. Kyoto R&D Center, Study Director — Clinical Development Department
Locations (3):
- Japan (3):
  - Sapporo, Hokkaido
  - Yokohama, Kanagawa
  - Nakano-Ku, Tokyo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 106 sites in Japan from September 2013 to Jully 2015
Period: Overall Study
Arm/Group | ASP2151(200 mg) | ASP2151(400mg) | Valaciclovir
Started | 252 | 250 | 249
Full Analysis Set Included | 247 | 243 | 245
Full Analysis Set Excluded | 5 | 7 | 4
Reason FAS Excluding 1 (Subjects who are found not to have herpes zoster) | 5 | 5 | 4
Reason FAS Excluding 2 (Those who have not received any dose of the study drug after randomization.) | 0 | 1 | 0
Reason FAS Excluding 3 (Those who have no efficacy assessment data after study drug administration.) | 0 | 1 | 0
Completed | 209 | 193 | 206
Not Completed | 43 | 57 | 43
Not completed — Adverse Event | 1 | 3 | 2
Not completed — Lack of Efficacy | 5 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Physician Decision | 0 | 2 | 3
Not completed — Protocol Violation | 16 | 23 | 16
Not completed — Withdrawal by Subject | 7 | 7 | 5
Not completed — Clinical laboratory value | 2 | 6 | 6
Not completed — Platelet count below on day1 or 4 | 11 | 15 | 11

BASELINE CHARACTERISTICS:
Population: The full analysis set(FAS).The FAS was defined as patients who were diagnosed with herpes zoster at the time of case registration, who subsequently received the study drugs, and had any efficacy variable measured.
Groups:
- Total: Total of all reporting groups
Arm/Group | ASP2151(200 mg) | ASP2151(400mg) | Valaciclovir | Total
Number analyzed (Participants) | 247 | 243 | 245 | 735
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 178 | 174 | 178 | 530
  >=65 years | 69 | 69 | 67 | 205
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (16.3) | 53.0 (16.2) | 52.2 (15.8) | 52.39 (16.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 134 | 144 | 146 | 424
  Male | 113 | 99 | 99 | 311
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 247 | 243 | 245 | 735
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 247 | 243 | 245 | 735
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 247 | 243 | 245 | 735
Time from onset of rash to the first dose [Count of Participants; unit: Participants]
  within 24 hours | 53 | 56 | 45 | 154
  over 24 hours, within 48 hours | 92 | 98 | 91 | 281
  over 48 hours, within 72 hours | 102 | 89 | 109 | 300

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants Achieving Cessation of New Lesion Formation by Day 4 of Study Treatment
Description: The investigator assessed the Number of rashes (erythemas/papulae and vesicles/pustules). The "new lesion formation" was defined as the state in which the number of rashes is increasing.
Time Frame: 4days
Population: as for baseline characteristics
Measure: Number; unit: percentage of Participants
Arm/Group | ASP2151(200 mg) | ASP2151(400mg) | Valaciclovir
Number analyzed (Participants) | 247 | 243 | 245
percentage of Participants | 69.6 | 81.1 | 75.1
Statistical Analysis 1: Comparison: ASP2151(400mg) vs Valaciclovir; The non-inferiority of each ASP2151 dose level versus valaciclovir was assessed stepwise using a closed testing procedure.First step analysis was performed in the ASP2151(400mg) once daily; Test type: Non-Inferiority — Wherein the non-inferiority margin was set at 10%. If the one-sided P-value was less than 0.025 between the ASP2151(400mg) once daily and the valaciclovir 1000 mg three times daily, non-inferiority of ASP2151 to valaciclovir was assumed; p = 0.00000241, Modified Farrington-Manning test
Statistical Analysis 2: Comparison: ASP2151(200 mg) vs Valaciclovir; The analysis was performed in the ASP2151(200 mg) once daily only when non-inferiority of the ASP2151(400 mg) 0nce daily to valaciclovir 1000 mg three times daily was assumed; Test type: Non-Inferiority — Wherein the non-inferiority margin was set at 10%. If the one-sided P-value was less than 0.025 between the ASP2151(200mg) once daily and the valaciclovir 1000 mg three times daily, non-inferiority of ASP2151 to valaciclovir was assumed; p = 0.0688, Modified Farrington-Manning test

2. Secondary Outcome: Time to Cessation of New Lesion Formation
Description: as for outcome 1
Time Frame: 29days
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | ASP2151(200 mg) | ASP2151(400mg) | Valaciclovir
Number analyzed (Participants) | 247 | 243 | 245
days | 4 [3 to 5] | 4 [3 to 4] | 4 [3 to 4]

3. Secondary Outcome: Time to Complete Crusting
Description: We defined the following state as "Complete crusting".
  1. A condition where all lesions of erythemas/papulae, vesicles/pustules, and erosions/ulcers have disappeared, and all rashes are crusted (epithelialization of the base of crusts is not required).
  2. In subjects with no formation of vesicles or pustules, a condition where all lesions of erythemas/papulae have disappeared.
Time Frame: 29days
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | ASP2151(200 mg) | ASP2151(400mg) | Valaciclovir
Number analyzed (Participants) | 247 | 243 | 245
days | 8 [6 to 11] | 9 [7 to 11] | 8 [7 to 11]

4. Secondary Outcome: Time to Healing
Description: We defined the following state as "Healing".
  1. A condition where all lesions of erythemas/papulae, vesicles/pustules, and erosions/ulcers have disappeared, and complete disappearance of crusts or complete epithelialization of the base of crusts are considered to have been achieved.
  2. In subjects with no formation of vesicles or pustules, a condition where all lesions of erythemas/papulae have disappeared
Time Frame: 29days
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | ASP2151(200 mg) | ASP2151(400mg) | Valaciclovir
Number analyzed (Participants) | 247 | 243 | 245
days | 11 [8 to 15] | 11 [8 to 15] | 11 [8 to 16]

5. Secondary Outcome: Time to Pain Resolution
Description: Investigators assessed the pain using NRS. The date of pain resolution is defined as the first day when all NRS scores are rated as 2 or less, and such scores are continuously observed until Day 92 or discontinuation visit.
Time Frame: 29days
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | ASP2151(200 mg) | ASP2151(400mg) | Valaciclovir
Number analyzed (Participants) | 247 | 243 | 245
days | 9 [5 to 19] | 10 [5 to 19] | 10 [5 to 19]

6. Secondary Outcome: Time to Virus Disappearance
Description: Virus desiappearance was defined as the participants who who reached virus-negative status according to the virus isolation and culture assay or whose samples were not available because of complete crusting or healing
Time Frame: 29days
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | ASP2151(200 mg) | ASP2151(400mg) | Valaciclovir
Number analyzed (Participants) | 247 | 243 | 245
days | 4 [4 to 8] | 5 [4 to 10] | 4 [3 to 9]

ADVERSE EVENTS:
Time Frame: 92 days
Description: Participant who has not received any study drug after randomization excluded from the Number participants at Risk
Arm/Group | ASP2151(200 mg) | ASP2151(400mg) | Valaciclovir
All-Cause Mortality (participants affected / at risk) | 0/252 | 0/249 | 0/249
Serious Adverse Events (participants affected / at risk) | 1/252 | 1/249 | 3/249
Other Adverse Events (participants affected / at risk) | 62/252 | 64/249 | 65/249
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ASP2151(200 mg) (N=252) | ASP2151(400mg) (N=249) | Valaciclovir (N=249)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 | 0
Infectious mononucleosis (Infections and infestations) | 0 | 1 (1) | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1 (1)
Embolic cerebral infarction (Nervous system disorders) | 0 | 0 | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ASP2151(200 mg) (N=252) | ASP2151(400mg) (N=249) | Valaciclovir (N=249)
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 5
Stomatitis (Gastrointestinal disorders) | 1 | 7 | 0
Folliculitis (Infections and infestations) | 5 | 0 | 5
Nasopharyngitis (Infections and infestations) | 19 | 22 | 17
Beta-N-acetyl-D-glucosaminidase increased (Investigations) | 7 | 11 | 8
Fibrin degradation products increased (Investigations) | 7 | 9 | 10
Glucose urine present (Investigations) | 3 | 3 | 5
Protein urine present (Investigations) | 2 | 5 | 5
Alpha 1 microglobulin increased (Investigations) | 11 | 9 | 10
Headache (Nervous system disorders) | 9 | 2 | 7
Dermatitis contact (Skin and subcutaneous tissue disorders) | 4 | 5 | 5
Eczema (Skin and subcutaneous tissue disorders) | 7 | 3 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes